CLINICAL TRIAL: NCT06637969
Title: Effects of Mindfulness-based Interventions on Psychophysiological Recovery and Physical Functioning in Patients After Coronary Heart Surgery
Brief Title: Mindfulness-based Interventions on Psychophysiological Recovery and Physical Functioning After Coronary Heart Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D528
Record Dates: First submitted 2024-08-23; First posted 2024-10-15 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Coronary Heart Disease; Mindfulness; Recovery, Psychological; Physical Functioning
Keywords: coronary heart disease surgery, mindfulness
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mindfulness-based (Experimental): The experimental group was also provided with a total of 30 minutes of mindfulness training once a day for seven consecutive days. The content included mindful breathing awareness for 8 minutes while resting and lying in bed, 10 minutes of mindfulness meditation, 12 minutes of mindfulness body scanning, and 10 minutes of mindful walking and breathing. The control group The group received routine care, and a pre-test was conducted before the implementation of the interventional measures (from 7 pm to 9 pm the day before the operation), and a post-test was conducted after the seven-day intervention (from 7 pm to 9 pm on the seventh day of the interventional treatment). Comparison between the experimental group and the control group group differences
  Interventions: Behavioral: mindfulness-based

INTERVENTIONS:
Behavioral: mindfulness-based — The experimental group was also provided with a total of 30 minutes of mindfulness training once a day for seven consecutive days. The content included mindful breathing awareness for 8 minutes while resting and lying in bed, 10 minutes of mindfulness meditation, 12 minutes of mindfulness body scanning, and 10 minutes of mindful walking and breathing. The control group The group received routine care, and a pre-test was conducted before the implementation of the interventional measures (from 7 pm to 9 pm the day before the operation), and a post-test was conducted after the seven-day intervention (from 7 pm to 9 pm on the seventh day of the interventional treatment). Comparison between the experimental group and the control group group differences

SUMMARY:
The purpose of this study is to explore the effect of mindfulness on the physical and mental recovery and physical function of patients after coronary heart surgery. Methods: Convenience sampling was adopted, and patients in the cardiology ward of a northern medical center were selected as the research subjects. Eligible subjects were assigned to the experimental group (mindfulness treatment) and the routine care group. The subjects were tested on the day before surgery and on the seventh day after intervention. Physical and mental recovery (awareness of inner feelings, anxiety, depression, sleep quality, pain) and physical function (vital capacity, cardiorespiratory endurance, dyspnea after exercise) were measured,

DETAILED DESCRIPTION:
Background: If patients with coronary heart disease are not properly controlled and treated, it is not only easy for the disease to relapse and cause angina pectoris, which will prevent the heart from receiving sufficient blood and oxygen supply, leading to an increase in the severity of the disease, and may lead to coronary artery bypass surgery, but postoperative complications may occur. Due to reduced respiratory muscle vitality, chest wound pain caused by median sternotomy surgery, and bed rest, resulting in incomplete lung expansion or lung collapse, discomfort due to physiological symptoms, and fear of life-threatening disease, and the risk of disease The uncertainty of treatment causes patients to have negative emotions of anxiety and depression, affecting their sleep quality. Purpose: The purpose of this study is to explore the effect of mindfulness on the physical and mental recovery and physical function of patients after coronary heart surgery. Methods: Convenience sampling was adopted, and patients in the cardiology ward of a northern medical center were selected as the research subjects. Eligible subjects were assigned to the experimental group (mindfulness treatment) and the routine care group. The subjects were tested on the day before surgery and on the seventh day after intervention. Physical and mental recovery (awareness of inner feelings, anxiety, depression, sleep quality, pain) and physical function (vital capacity, cardiorespiratory endurance, dyspnea after exercise) were measured, and the secondary measurement data were statistically analyzed using SPSS 29.0 for Windows software suite. Compare the differences between the two groups in physical and mental recovery and physical function.

ELIGIBILITY:
Inclusion Criteria 18Aged Patients who are hospitalized and expected to undergo coronary artery bypass surgery Those who can cooperate with regular use of induction spirometry Exclusion Criteria major mental illnesses cognitive impairment long-term bed rest mobility difficulties have deformities of the mouth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Multidimensional assessment of interoceptive awareness | one year
  The inner feeling awareness scale covers eight factors: attention, non-distraction, non-worry, concentration adjustment, emotional awareness, self-regulation, body listening, and trust, with a total of 32 questions. The questionnaire is scored on a scale of 0-5 based on the response content, with higher scores indicating more positive inner feeling awareness.

SECONDARY OUTCOMES:
Incentive Spirometer | one year
  When the first ball is sucked up and reaches the top for one second, the lung ventilation volume is 600ml/second. When the second ball is sucked up and reaches the top, the lung ventilation volume is 900ml/second. When starting and reaching the peak, the lung ventilation volume is 1200ml/second.
Verran and Snyder Halpen Sleep scale | one year
  The sleep quality referred to in this study uses the Chinese version of the Weixin Sleep Scale compiled by Lin Xiaoling and Cai Xinling to evaluate the subjective feelings of sleep last night (from 10 clock last night to 8 clock in the morning). Its content covers sleep disturbance, sleep effectiveness and sleep supplementation There are three factors, a total of 15 questions. The questionnaire is scored on a scale of 0-100 according to the answer content. The minimum score for each positive question is 0 points and the maximum score is 100 points. The total score is 0-1500 points. The higher the score, the better the sleep quality.
Hospital Anxiety and Depression Scale | one year
  This scale was developed by Zigmond and Snaith in 1983 to measure patients; anxiety and depression. It has 14 questions in total. The higher the score, the higher the degree of anxiety or depression. The odd-numbered questions assess anxiety, and the even-numbered questions assess depression. A score of 0-7 indicates no anxiety or depression, a score of 8-10 indicates a borderline case, and a score of 11-21 indicates anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Taiwan Presbyterian Church Mackay Medical Foundation Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No